CLINICAL TRIAL: NCT01336153
Title: Clinical Study to Investigate the Safety and Efficacy of MLC601 in 150 Iranian Patients After Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Mostafa Ghanei, Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN89-01-117-7548
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2010-12

CONDITIONS: Stroke
Keywords: Safety; Efficacy; MLC601; motor recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MLC601 (Experimental): MLC601 (NeuroAideTM) is a TCM which is used extensively in China to improve recovery after stroke. It combines several herbal and animal components.
  Interventions: Drug: MLC601
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLC601 — group A (100 patients; NeuroAid 400mg, 4 capsules 3 times daily) or for 3 month
  Arms: MLC601
Drug: Placebo — group B (50 patients; placebo, 4 capsules 3 times daily) for 3 months
  Arms: Placebo

SUMMARY:
To investigate the safety and efficacy of MLC601 (NeuroAideTM) as a Traditional Chinese Medicine on motor recovery after ischemic stroke.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled clinical trial study on 150 patients with a recent (less than 3 month) ischemic stroke. All patients will give either MLC601 (100 patients) or placebo (50 patients), 4 capsules 3 times a day, as an add-on to standard medication of post stroke for 3 months. Motor improvement will be monitored using Fugl-Meyer Assessment FMA.

ELIGIBILITY:
Inclusion Criteria:

* age between 30-72 yars,
* < one month after stroke,
* ischemic cerebral stroke,
* signed informed consent form.

Exclusion Criteria:

* treatment with thrombolytic after stoke,
* ischemic stroke combined with hemorrhage, severe renal or liver failure, dementia, psychosis and history of seizure disorder, history of previous stroke, and hemoglobin level less than 10mg/dl on admission.

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Investigate the Safety and Efficacy of MLC601 | 18 months
  Patients showed a good tolerability to treatment and adverse events were mild and transient.

SECONDARY OUTCOMES:
Motor recovery of MLC601 in 150 Iranian Patients after Stroke | 18 months
  Repeated measured analysis showed statistically difference in Fugl-Meyer Assessment FMA score during 12 months between two groups